CLINICAL TRIAL: NCT04512495
Title: Circulating " Cancer Cells / Macrophage " HYbrid Cells in Patients With Sarcoma?
Acronym: SAMHY SARCOME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20 SARC 04
Record Dates: First submitted 2020-08-07; First posted 2020-08-13 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Sarcoma
Keywords: Leiomyosarcoma; Dedifferentiated liposarcoma; Myxoid liposarcoma; Synovialosarcoma; Osteosarcoma; Ewing's sarcoma; Cancer cell/macrophage hybrid cells; Hybrid cells
MeSH Terms: conditions — Sarcoma; Leiomyosarcoma; Liposarcoma; Liposarcoma, Myxoid; Sarcoma, Synovial; Osteosarcoma; Sarcoma, Ewing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with sarcoma (Other)
  Interventions: Other: Blood samples will be collected at two times :

INTERVENTIONS:
Other: Blood samples will be collected at two times : — * at Baseline,
  * after surgery or at the time of post-chemotherapy evaluation.

SUMMARY:
Pilot, prospective, monocentric study aimed at evaluating the rate of patients with circulating "cancer cell/macrophage" hybrid cells in the peripheral blood.

The study will be conducted on a population of patients with sarcoma and treated in the context of routine care.

For each included patient, blood samples will be collected during baseline visit and after the initiation therapy.

At the end of the 2nd blood collection, the patient will have completed his participation in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with one of the following subtypes of soft tissue or bone sarcomas: leiomyosarcoma, dedifferentiated liposarcoma, myxoid liposarcoma, synovialosarcoma, osteosarcoma, Ewing's sarcoma.
2. Diagnosis of sarcoma histologically confirmed by the RRePS network (Réseau de Référence en Pathologie des Sarcomes et des Viscères)
3. Age ≥ 18 years old.
4. Localized or metastatic disease or recurrent disease.
5. Patient who has not yet initiated specific treatment for sarcoma.
6. Patient affiliated to a Social Health Insurance in France.
7. Patient having signed informed consent prior to inclusion in the study and prior to any specific study procedures.

Exclusion Criteria:

1. Patient with any other histological subtype of sarcoma, including pleomorphic sarcoma.
2. Associated pathology(s) that may prevent the proper conduct of the procedure under consideration.
3. Pregnant or breastfeeding woman.
4. Any psychological, family, geographical or sociological condition that prevents compliance with the medical follow-up and/or procedures of the study protocol.
5. Patient who has forfeited his/her freedom by administrative or legal award or who is under legal protection (curatorship and guardianship, protection of justice).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
Rate of patients with "cancer cell / macrophage" hybrid cells in peripheral blood. | 6 months after the end of inclusions

SECONDARY OUTCOMES:
Quantification of circulating hybrid cells in peripheral blood by automatic measurement (Cell Counter Corning) and expressed in number of cells / millilitre of blood. | 6 months after the end of inclusions

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse, France